CLINICAL TRIAL: NCT06578078
Title: A Randomized Clinical Trial to Define the Best Strategy for the Management of Heart Failure and Chronic Kidney Disease Among Elderly Patients With or at High Risk of hyperKalemia in Span by Optimizing the Use of RAASi With SZC
Brief Title: A Clinical Trial to Define the Best Strategy for the Management of Heart Failure in Elderly Patients
Acronym: SENEKA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENEKA; 2024-513971-42-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Chronic Kidney Diseases
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Intervention Model Description: This is a randomised clinical trial, multicentre, open label, of RAASi associated with SZC versus modification of RAASi without added chelator in patients over 70 years of age, who after the stabilization of an acute HF episode and comorbid CKD, have HK or are at high risk of developing HK.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SZC group (Experimental): Sodium zirconium cyclosilicate with standard of care treatment (RAASi therapy)
  Interventions: Drug: Sodium Zirconium Cyclosilicate
- Control group (Active Comparator): Standard of care treatment (RAASi therapy) without Sodium zirconium cyclosilicate
  Interventions: Drug: Standard of care treatment (RAASi therapy)

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate — Use of sodium zirconium cyclosilicate to optimize RAASi therapy, through up-titration of ACEi, ARB, ARNI or MRA therapy according to clinical guidelines
  Other Names: Lokelma
  Arms: SZC group
Drug: Standard of care treatment (RAASi therapy) — Standard of care treatment (RAASi therapy) without use of sodium zirconium cyclosilicate
  Arms: Control group

SUMMARY:
Heart failure (HF) and Chronic Kidney Disease (CKD) patients are frequently not administered renin-angiotensin aldosterone system inhibitor (RAASi) therapies at recommended doses due to hyperkalaemia, despite proven mortality and morbidity benefits. Sodium zirconium cyclosilicate (SZC) is a nonabsorbed potassium binder proven to lower serum potassium (S-K) and maintain normokalaemia. The purpose is to assess if a treatment regimen containing SZC will allow RAASi therapies to be optimized to target doses in patients with heart failure, chronic kidney disease and elevated serum potassium or at risk of developing elevated serum potassium.

DETAILED DESCRIPTION:
This is a randomized clinical trial, multicentre, parallel group, open label, to evaluate the use of sodium zirconium cyclosilicate (SZC) to optimize RAASi therapy in patients with heart failure and chronic kidney disease, through up-titration of ACEi, ARB, ARNI or MRA therapy according to clinical guidelines (1), without inducing clinically significant hyperkalemia. Eligible subjects will have been admitted to hospital because of an HF (NYHA I- III) decompensation, will have required intravenous diuretics and will have had mild hyperkalaemic values that needed stabilization or be at risk of developing hyperkalaemia. Subjects will be randomised in a 1:1 ratio to receive SZC or none (standard of care treatment without potassium binders) for 3 months while optimizing RAASi therapies according to the European Society of Cardiology (ESC) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Provision of informed consent form prior to any study specific procedures, sampling and analysis.
* Individuals must be ≥ 70 years of age at the time of signing the informed consent form.
* Individuals must have a confirmed diagnosis of Heart Failure (HF) according to clinical practice guidelines NYHA functional class I-III (with HFrEF or HFpEF).
* Individuals must have previously been admitted to hospital due to HF decompensation requiring intravenous diuretics.
* Individuals must have been stabilised for at least 24-48h of their HF decompensation before randomisation.
* Individuals must have a confirmed diagnosis of Chronic Kidney Disease defined as a renal impairment of eGFR less than 60ml/min/1.73 m2.
* Individuals receiving background standard of care for HF and treated according to international guidelines. Specific treatment should include RAASi and/or MRA treatment and at least should have been stable for ≥ 4 weeks at maximum tolerated doses.
* Patients on RAASi blocker treatment with less than or equal to 75% of the maximum recommended dose.
* Hyperkalemic patients (sK+ 5.1-5.9 mmol/L at screening / study enrolment) or Normokalemic patients at risk of developing HK defining as having a history of hyperkalaemia (sK+ >5.0 mEq/L) within the prior 24 months and sK+ ≥4.5 mEq/L ≤ 5.1 mEq/L at inclusion

Exclusion Criteria:

* Limited life expectancy (less than 1 year) according to clinician's criteria, such as but not limited to malignancy, with life expectancy of less than 2 years based on investigator's clinical judgement.
* sK >6 mEq/litre or <4.5mEq/litre or history of hypokalemic episodes (S-K<3.5 mEq/L) during the last year.
* Patients on haemodialysis or haemofiltration
* NYHA functional class IV
* Patients undergoing treatment with potassium binders.
* Active tumour undergoing chemotherapy or metastasis or malignancy requiring treatment.
* Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled by medication are permitted.
* QTc(f) > 550 msec.
* History of QT prolongation associated with other medications that required discontinuation of that medication.
* Congenital long QT syndrome.
* Prior history of hypersensitivity to a RAAS blocker drug, including but not limited to development of angioedema, icterus, hepatitis, or neutropenia or thrombocytopenia requiring treatment modification. Addison's disease or other causes of hypoaldosteronism.
* Patients with a known hypersensitivity to SZC or any of the excipients of the product.
* Individuals treated with potassium binding resins such as sodium polystyrene sulfonate (SPS, e.g. Kayexalate®) or calcium polystyrene sulfonate (CPS; e.g. Resonium®) or the cation exchange polymer, patiromer sorbitex calcium (Veltassa®) within 7 days prior to the first dose of study drug.
* Treated with potassium supplements within 7 days prior to randomization. 15. Positive hepatitis C antibody hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening.
* Known to have tested positive for human immunodeficiency virus.
* Known history of drug or alcohol abuse within 3 year of screening.
* Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site).
* Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions and requirements.
* Previous enrolment in the present study.
* Participation in another clinical study with an investigational product during the last 3 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients increasing at least 25% of the target doses of RAASi since the screening visit (V0) to 3 months after study inclusion (V9) | Through study completion, an average of 3 months
  To compare the number of patients achieving an increase of at least 25% of RAASi according to guideline-recommended target doses, in the arm treated with Lokelma plus RAASi versus the arm treated with RAASi without K+ binder, at 3 months after study inclusion.

SECONDARY OUTCOMES:
Number of patients achieving at least 50% of the target doses of RAASi since the screening visit (V0) to 3 months after study inclusion (V9) | Through study completion, an average of 3 months
  To assess the number of patients achieving at least 50% of the target dose of RAASi recommended in the guidelines.
Number of patients increasing 50% of RAASi doses since the screening visit (V0) to 3 months after study inclusion (V9) | Through study completion, an average of 3 months
  To assess the number of patients achieving at least 50% of the target dose of RAASi recommended in the guidelines.

OTHER OUTCOMES:
Number of patients achieving at least 50% of the target doses of MRA since the screening visit (V0) to 3 months after study inclusion (V9) | Through study completion, an average of 3 months
  To assess the number of patients that achieve at least 50% of the target dose recommended in guidelines of Mineralocorticoid receptor antagonist (MRA).
Number of patients increasing 50% of MRA doses since the screening visit (V0) to 3 months after study inclusion (V9) | Through study completion, an average of 3 months
  To assess the number of patients that achieve at least 50% of the target dose recommended in guidelines of Mineralocorticoid receptor antagonist (MRA)
Number of patients achieving at least 50% of the target doses of MRA and RAASi since the screening visit (V0) to 3 months after study inclusion (V9) | Through study completion, an average of 3 months
  To analyse the number of patients achieving at least 50% of the recommended target dose of MRA and achieving at least 50% of the guidelines recommended target dose of RAASi
Number of patients increasing 50% of MRA and RAASi doses since the screening visit (V0) to 3 months after study inclusion (V9) | Through study completion, an average of 3 months
  To analyse the number of patients achieving at least 50% of the recommended target dose of MRA and achieving at least 50% of the guidelines recommended target dose of RAASi
Number of patients achieving the target doses of RAASi since the screening visit (V0) to 3 months after study inclusion (V9) | Through study completion, an average of 3 months
  To evaluate the number of patients achieving the target dose recommended in guidelines of RAASi.
Proportion of patients in each group requiring a down titration of RAASi and/or MRA over the study period | Through study completion, an average of 3 months
  To evaluate the number of patients requiring down titration and discontinuation of RAASi and/or MRA during the study
Proportion of patients in each group requiring up titration of RAASi and/or MRA following down titration of RAASi and/or MRA | Through study completion, an average of 3 months
  To evaluate the number of patients requiring down titration and discontinuation of RAASi and/or MRA during the study
Proportion of patients in each group requiring discontinuation of RAASi and/or MRA over the study period. | Through study completion, an average of 3 months
  To evaluate the number of patients requiring down titration and discontinuation of RAASi and/or MRA during the study
Number of patients achieving at least 50% of the target doses of RAASi since the screening visit (V0) to 1 month after study inclusion | Through study completion, an average of 3 months
  To analyse the number of patients achieving 50% of target doses recommended in guidelines of RAASi at 1 month after study inclusion
Number of patients increasing 50% of RAASi doses since the screening visit (V0) to 1 month after study inclusion | Through study completion, an average of 3 months
  To analyse the number of patients achieving 50% of target doses recommended in guidelines of RAASi at 1 month after study inclusion
Number of patients achieving a decrease of at least 5% in NT-proBNP levels since the baseline visit (V1) to 3 months after study inclusion (V9). | Through study completion, an average of 3 months
  To determine surrogate short-term (90 days) efficacy objective of changes in biomarker levels (NT-proBNP and CA125) evaluated as a decrease of at least 5% from baseline to 3 months after study inclusion.
Mean Change in NT-proBNP levels since the baseline visit (V1) to 3 months after study inclusion (V9). | Through study completion, an average of 3 months
  To determine surrogate short-term (90 days) efficacy objective of changes in biomarker levels (NT-proBNP and CA125) evaluated as a decrease of at least 5% from baseline to 3 months after study inclusion.
Number of patients achieving a decrease of at least 5% in CA125 levels since the baseline visit (V1) to 3 months after study inclusion (V9). | Through study completion, an average of 3 months
  To determine surrogate short-term (90 days) efficacy objective of changes in biomarker levels (NT-proBNP and CA125) evaluated as a decrease of at least 5% from baseline to 3 months after study inclusion.
Mean Change in CA125 levels since the baseline visit (V1) to 3 months after study inclusion (V9). | Through study completion, an average of 3 months
  To determine surrogate short-term (90 days) efficacy objective of changes in biomarker levels (NT-proBNP and CA125) evaluated as a decrease of at least 5% from baseline to 3 months after study inclusion.
Mean change on Systolic arterial blood pressure measurement from baseline visit (V1) to 3 months after study inclusion (V9). | Through study completion, an average of 3 months
  To explore changes in systolic arterial blood pressure at baseline and 3 months after study inclusion.
Mean change from baseline visit (V1) measured at 3 months after study inclusion (V9) in the overall summary score of KKCQ, as a specific HF patient reported outcome questionnaire. | Through study completion, an average of 3 months
  To explore the effect of treatment with SZC versus none on Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score.
To determine the change in renal function the Mean Change in UACR and Mean change in HCO3 will be calculated between baseline visit (V1) and 3 months after study inclusion (V9) | Through study completion, an average of 3 months
  To evaluate changes in renal function at baseline and 3 months after study inclusion between both groups
Number of patients decreasing at least 40% the eGFR since the screening visit (V0) to 3 months after study inclusion (V9). | Through study completion, an average of 3 months
  To analyse the number of patients that decrease at least 40% in estimated glomerular filtration rate (eGFR) by the CDK-EPI formula.
Mean change from baseline visit (V1) measured at 3 months after study inclusion (V9) in the overall summary score of KDQoL, as a specific CKD patient reported outcome questionnaire. | Through study completion, an average of 3 months
  To explore the effect of treatment with SZC versus none on the Kidney Disease Questionnaire of life (KDQoL) Overall Summary Score.
Number of visits for HF/HK/impaired renal function/hypertension or hyperkalemia diagnosed in the outpatient clinic. | Through study completion, an average of 3 months
  To determine the number of visits to the emergency department for HF/HK/impaired renal function/hypertension (defined as BP over 200 and/or 100 mmHg) and hyperkalemia diagnosed in the outpatient clinic.
Proportion of patients requiring hospitalization for HF/HK/impaired renal function over the study period. | Through study completion, an average of 3 months
  To analyse the number of admissions for HF/HK/impaired renal function.
Mean number of hospitalizations per patient for HF/HK/impaired renal function over the study period. | Through study completion, an average of 3 months
  To analyse the number of admissions for HF/HK/impaired renal function.
Proportion of patients presenting at least one clinical event over the study period | Through study completion, an average of 3 months
  To evaluate in both experimental groups the combined endpoint of visits to the emergency department or admission for HF/HK/impaired renal function or decrease of at least 40% in estimated glomerular filtration rate (eGFR) by the CDK-EPI formula or death from cardiovascular causes.
Proportion of patients presenting more than one clinical event over the study period | Through study completion, an average of 3 months
  To evaluate in both experimental groups the combined endpoint of visits to the emergency department or admission for HF/HK/impaired renal function or decrease of at least 40% in estimated glomerular filtration rate (eGFR) by the CDK-EPI formula or death from cardiovascular causes.
Proportion of patients presenting all clinical events over the study period | Through study completion, an average of 3 months
  To evaluate in both experimental groups the combined endpoint of visits to the emergency department or admission for HF/HK/impaired renal function or decrease of at least 40% in estimated glomerular filtration rate (eGFR) by the CDK-EPI formula or death from cardiovascular causes.
Percentage of patients treated with and without sodium-glucose cotransporter-2 (SGLT2) inhibitors over the study period in both arms | Through study completion, an average of 3 months
  To analyse the percentage of patients with HF treated with and without sodium-glucose cotransporter-2 (SGLT2) inhibitors.
Mean Change in Mg levels since the baseline visit (V1) to 3 months after study inclusion (V9). | Through study completion, an average of 3 months
  To explore changes in Mg levels at baseline and 3 months after study inclusion.
Proportion of patients presenting each clinical outcome over the study period: Adverse events, Serious adverse events, Changes in clinical laboratory parameters, Changes in vital signs and ECGs | Through study completion, an average of 3 months
  To evaluate the safety and tolerability of SZC in this patient population.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Nuestra Señora del Perpétuo Socorro, Albacete
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No